CLINICAL TRIAL: NCT01982084
Title: Attitudes to Immunisation Against Group B Streptococcus During Pregnancy in England and Scotland
Brief Title: Group B Streptococcus: Attitudes to Immunisation in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: St George's, University of London (Other); University College, London (Other); Imperial College London (Other); Royal Infirmary of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: OVG2013/06
Record Dates: First submitted 2013-10-10; First posted 2013-11-13 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Immunisation During Pregnancy; Group B Streptococcus
Keywords: Group B streptococcus; Immunisation; Pregnancy; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Group B Streptococcus (GBS) is the commonest cause of severe infection and meningitis in babies under 3 months in the United Kingdom (UK). About one in ten babies with GBS infection die and half of babies with GBS meningitis are left with long term problems with their development.

Vaccinating pregnant women against GBS in order to protect their newborn babies is a promising area of research.However, many women are reluctant to accept vaccination during pregnancy for fear it will harm their unborn child and there is often a lack of understanding of both the vaccine and the condition it aims to prevent. Nevertheless, the recent positive experience of immunisation against pertussis in the United Kingdom, suggest that antenatal immunisation can be acceptable.

Previous research has shown that advice from maternity healthcare professionals regarding vaccination is highly valued by pregnant women so it is also important to explore the attitudes and opinions of this group.

The objective of this study is to assess the knowledge and attitudes of pregnant women and maternity healthcare professionals in England and Scotland regarding GBS disease and the acceptability of a potential vaccine.

There are two parts to this study. The first part will invite pregnant women, maternity healthcare professionals and parents who have had a child affected by GBS disease to take part in either a focus group or an individual interview.

This will allow for an in-depth exploration of the participants thoughts and opinions about GBS and vaccination in pregnancy. This part of the study will take place at the Oxford site only. The results will guide the development of a self completed, paper questionnaire which will be distributed to a wider range of pregnant women and maternity healthcare professionals across four different study sites.

This study has been funded by Meningitis UK. Additional collaborators to those listed include the charity Group B Strep Support.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years and above who have not previously had a child with GBS disease and are willing and able to give written, informed consent and are able to read and speak English. OR
* Obstetricians (including consultants and trainees) or midwives working at one of the study site who are willing and able to give written, informed consent OR
* Parents (mothers or fathers) of children who have had GBS disease (early or late onset), potentially including parents of children who have died from GBS disease who are willing and able to given written, informed consent Able to read and speak English

Exclusion Criteria:

* The inclusion criteria are not met
* Volunteer is part of the study team at any of the study sites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women aged 18 years and over of any gestation receiving antenatal care in the Oxford area (part one and two) or within Imperial college and St Georges's NHS trusts in London and Edinburgh Royal infirmary (part two).
  Maternity healthcare professionals (midwives and doctors)working in the above areas.
  Parents who have had a child with Group B streptococcal disease (part one only).
Sampling Method: Non-Probability Sample
Enrollment: 758 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03-29 (Actual)

PRIMARY OUTCOMES:
The attitudes of pregnant women and maternity healthcare professionals towards vaccination against Group B streptococcus in pregnancy | Single timepoint at interview or focus group lasting on average 1-2 hours
  The attitude of pregnant women and maternity healthcare professionals will be measured using their responses to questions asked during interviews or focus groups

OTHER OUTCOMES:
Attitudes of pregnant women to participating in a clinical trial of a GBS vaccine | Single time point at interview or focus group lasting on average 1-2 hours
  The attitudes of pregnant women to participating in a clinical trial of a GBS vaccine and the potential barriers and motivations to participation and how these could be addressed will be measured using the responses to questions asked during hte interview/focus group sessions

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Snape, MBBS FRCPCH, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - Edinburgh Royal Infirmary, Edinburgh
  - Imperial College London, London
  - St Georges University of London, London
  - Oxford Vaccine Group, University of Oxford, Oxford

REFERENCES:
- [Result] McQuaid F, Pask S, Locock L, Davis E, Stevens Z, Plumb J, Snape MD. Attitudes towards antenatal vaccination, Group B streptococcus and participation in clinical trials: Insights from focus groups and interviews of parents and healthcare professionals. Vaccine. 2016 Jul 25;34(34):4056-61. doi: 10.1016/j.vaccine.2016.06.024. Epub 2016 Jun 16. PMID 27318418
- [Result] McQuaid F, Jones C, Stevens Z, Meddaugh G, O'Sullivan C, Donaldson B, Hughes R, Ford C, Finn A, Faust SN, Gbesemete D, Bedford H, Hughes S, Varghese AS, Heath PT, Snape MD. Antenatal vaccination against Group B streptococcus: attitudes of pregnant women and healthcare professionals in the UK towards participation in clinical trials and routine implementation. Acta Obstet Gynecol Scand. 2018 Mar;97(3):330-340. doi: 10.1111/aogs.13288. Epub 2018 Jan 19. PMID 29292509